CLINICAL TRIAL: NCT05417607
Title: Sub-study: Feasibility Trial of Adapted ESDM-informed Caregiver Coaching Delivered Remotely for Children With ASD and ADHD
Brief Title: A+ Treatment/Feasibility of Adapted ESDM-informed Caregiver Coaching Delivered Remotely for Children With ASD (Autism Spectrum Disorder) and ADHD (Attention Deficit Hyperactivity Disorder)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00085179_1
Record Dates: First submitted 2022-05-25; First posted 2022-06-14 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder; Adhd
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Feasibility trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A+ Treatment/Feasibility participants (Other): Total participation is expected to require a maximum of 20 weeks (plus optional remote follow-up at 16 week). Diagnostic/screening visits occur between 1 and 6 weeks prior to baseline and start of coaching. ESDM-informed parent coaching (~1 hour sessions) is delivered remotely (through telehealth) with a study clinician for 8 weeks and strategies are implemented within the child's typical daily routines by the caregiver. No medication is provided by the study team. Data is collected weekly and final assessment will be obtained at 16 weeks after baseline.
  Interventions: Behavioral: P-ESDM informed caregiver coaching

INTERVENTIONS:
Behavioral: P-ESDM informed caregiver coaching — Caregiver coaching informed by P-ESDM done remotely (via telehealth)

SUMMARY:
This study will evaluate the feasibility of adapted ESDM-informed caregiver coaching in children with comorbid ASD and ADHD, who are between 36 and <132 months of age. There will be no study provided medication treatment in this study. Children will either be on ADHD medication prescribed by their own personal provider or will not be taking any ADHD medication (this will be documented by the study). The provided behavioral treatment will be eight ~60-minute sessions in ESDM-informed caregiver coaching delivered remotely through telehealth, for 8 consecutive weeks. The behavioral treatment is provided to children through Early Start Denver Model (ESDM)-informed caregiver coaching strategies, implemented within the child's typical daily routine by the caregiver.

DETAILED DESCRIPTION:
The overarching goal of A+ Treatment is to evaluate feasibility and gather pilot data of remotely-delivered ESDM informed caregiver coaching for children with ASD and ADHD which may inform future combination clinical trials (pharmacotherapy and behavioral intervention). Using an implementation science approach, the investigators will characterize the acceptability, appropriateness, feasibility and fidelity of remote behavioral intervention. Approximately 30-35 participants who are between 36 months and <132 months of age with comorbid ASD and ADHD will take part in this study, which includes parent coaching sessions completed remotely. Total participation is expected to require a maximum of 20 weeks, including optional remote follow-up at 16 weeks. The A+ Treatment diagnostic and screening visits will generally occur between 1 and 6 weeks prior to baseline. The provided behavioral treatment will be eight ~60-minute weekly sessions of ESDM-informed caregiver coaching delivered remotely through telehealth, for 8 consecutive weeks. Endpoint assessments will be completed after the final coaching visit. No medication will be provided by the study team. The final assessment will be obtained at 16 weeks after baseline.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a parent/guardian signed and dated informed consent form.
* Stated willingness of parent/guardian to comply with all study procedures and availability for the duration of the study.
* Child is between 36 months and <132 months of age at baseline.
* Child has a confirmed DSM-5 diagnosis of both ASD and ADHD, informed by results of assessments including: an ASD diagnostic assessment (Brief Observation of Symptoms of Autism [BOSA], Autism Diagnostic Observation Schedule, 2nd Edition [ADOS-2], or TELE-ASD-PEDS, and if applicable the Autism Diagnostic Interview - Revised [ADI-R]) and an ADHD diagnostic (a standardized ADHD Diagnostic Interview and the MINI psychiatric diagnostic interview).

Exclusion Criteria:

* If continuing psychotropic (CNS-active) medications, must not have been changed within 4 weeks prior to baseline.
* Significant visual, auditory or motor impairments that would preclude participation in ESDM-informed caregiver coaching or completion of key assessments.
* Inability of the caregiver participating in ESDM-informed caregiver coaching and responding to questionnaires to fluently speak English.
* Study clinician judgment that it is not in the best interests of the participant and/or the study for the child to participate (including presence of psychiatric conditions or psychiatric symptoms in addition to ASD and ADHD that in the opinion of the PI or based on senior clinical review, would confound assessments and/or affect participation in the study).

Ages: 36 Months to 131 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Franz, M.B., CH.B., Principal Investigator — Duke University; Geraldine Dawson, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Through NDAR (National Database for Autism Research), core assessment and diagnostic data that is de-identified, including Vineland data and autism assessments.
Supporting Information: Study Protocol
Time Frame: 1 year after publication of the results for each of the specific aims or 3 years after the statistical analyses are completed
Access Criteria: determined by committee of researchers/administrator at NDAR
URL: https://nda.nih.gov

RESULTS

PARTICIPANT FLOW:
Groups:
- A+ Treatment Caregiver-Child Dyads - Caregivers: Participants in this arm will be caregivers of children with ASD (Autism Spectrum Disorder) and/or ADHD (Attention Deficit Hyperactivity Disorder).
  Total participation is expected to require a maximum of 20 weeks (plus optional remote follow-up at 16 week). Diagnostic/screening visits occur between 1 and 6 weeks prior to baseline and start of coaching. Early Start Denver Model (ESDM)-informed parent coaching (~1 hour sessions) is delivered remotely (through telehealth) with a study clinician for 8 weeks and strategies are implemented within the child's typical daily routines by the caregiver. No medication is provided by the study team. Data is collected weekly and final assessment will be obtained at 16 weeks after baseline.
  P-ESDM informed caregiver coaching: Caregiver coaching informed by P-ESDM done remotely (via telehealth)
- A+ Treatment Caregiver-Child Dyads - Children: Participants in this arm will be children with ASD (Autism Spectrum Disorder) and/or ADHD (Attention Deficit Hyperactivity Disorder).
  Total participation is expected to require a maximum of 20 weeks (plus optional remote follow-up at 16 week). Diagnostic/screening visits occur between 1 and 6 weeks prior to baseline and start of coaching. Early Start Denver Model (ESDM)-informed parent coaching (~1 hour sessions) is delivered remotely (through telehealth) with a study clinician for 8 weeks and strategies are implemented within the child's typical daily routines by the caregiver. No medication is provided by the study team. Data is collected weekly and final assessment will be obtained at 16 weeks after baseline.
  P-ESDM informed caregiver coaching: Caregiver coaching informed by P-ESDM done remotely (via telehealth)
- A+ Treatment Staff: Participants in this arm will be staff who provide A+ Treatment Early Start Denver Model (ESDM)-informed coaching.
  Total participation is expected to require a maximum of 20 weeks (plus optional remote follow-up at 16 week). Diagnostic/screening visits occur between 1 and 6 weeks prior to baseline and start of coaching. Early Start Denver Model (ESDM)-informed parent coaching (~1 hour sessions) is delivered remotely (through telehealth) with a study clinician for 8 weeks and strategies are implemented within the child's typical daily routines by the caregiver. No medication is provided by the study team. Data is collected weekly and final assessment will be obtained at 16 weeks after baseline.
  P-ESDM informed caregiver coaching: Caregiver coaching informed by P-ESDM done remotely (via telehealth)
Period: Overall Study
Arm/Group | A+ Treatment Caregiver-Child Dyads - Caregivers | A+ Treatment Caregiver-Child Dyads - Children | A+ Treatment Staff
Started | 26 | 26 | 5
Completed | 24 | 24 | 5
Not Completed | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Data was not collected on Caregivers of Staff.
Groups:
- A+ Treatment Caregiver-Child Dyads - Caregivers: Participants in this arm will be caregivers of children with ASD and/or ADHD.
  Total participation is expected to require a maximum of 20 weeks (plus optional remote follow-up at 16 week). Diagnostic/screening visits occur between 1 and 6 weeks prior to baseline and start of coaching. Early Start Denver Model (ESDM)-informed parent coaching (~1 hour sessions) is delivered remotely (through telehealth) with a study clinician for 8 weeks and strategies are implemented within the child's typical daily routines by the caregiver. No medication is provided by the study team. Data is collected weekly and final assessment will be obtained at 16 weeks after baseline.
  P-ESDM informed caregiver coaching: Caregiver coaching informed by P-ESDM done remotely (via telehealth)
- A+ Treatment Caregiver-Child Dyads - Children: Participants in this arm will be children with ASD and/or ADHD.
  Total participation is expected to require a maximum of 20 weeks (plus optional remote follow-up at 16 week). Diagnostic/screening visits occur between 1 and 6 weeks prior to baseline and start of coaching. Early Start Denver Model (ESDM)-informed parent coaching (~1 hour sessions) is delivered remotely (through telehealth) with a study clinician for 8 weeks and strategies are implemented within the child's typical daily routines by the caregiver. No medication is provided by the study team. Data is collected weekly and final assessment will be obtained at 16 weeks after baseline.
  P-ESDM informed caregiver coaching: Caregiver coaching informed by P-ESDM done remotely (via telehealth)
- Total: Total of all reporting groups
Arm/Group | A+ Treatment Caregiver-Child Dyads - Caregivers | A+ Treatment Caregiver-Child Dyads - Children | A+ Treatment Staff | Total
Number analyzed (Participants) | 0 | 26 | 0 | 26
Age, Continuous [Mean (Standard Deviation); unit: months] |  | 103.4 (19.8) |  | 103.4 (19.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 6 |  | 6
  Male |  | 20 |  | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 1 |  | 1
  Not Hispanic or Latino |  | 25 |  | 25
  Unknown or Not Reported |  | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 |  | 0
  Asian |  | 0 |  | 0
  Native Hawaiian or Other Pacific Islander |  | 0 |  | 0
  Black or African American |  | 6 |  | 6
  White |  | 15 |  | 15
  More than one race |  | 5 |  | 5
  Unknown or Not Reported |  | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  | 26 |  | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Caregivers and Staff Who Completed Individual Qualitative Interviews to Assess the Acceptability, Appropriateness, and Feasibility of the Intervention
Description: Questions are tailored to stakeholder group and are informed by previous studies that have examined barriers and facilitators during the implementation of a new treatment approach. Interviews will be conducted after completing coaching sessions. Qualitative analysis will use an iterative coding and review process informed by grounded theory.
Time Frame: Week 9/Endpoint
Population: Caregivers and staff who completed the individual qualitative interviews. Caregivers responded to the questions for both themselves and their child.
Measure: Count of Participants; unit: Participants
Arm/Group | A+ Treatment Caregiver-Child Dyads - Caregivers | A+ Treatment Staff
Number analyzed (Participants) | 24 | 5
Participants | 24 | 5

2. Primary Outcome: Feasibility of Intervention (as Measured by Feasibility of Intervention Measure, FIM)
Description: The FIM is a four-item implementation outcome measure that measures the extent to which a new treatment, or an innovation, can be successfully used or carried out within a given agency or setting. Each item is rated on a 5-point ordinal scale from 1 (completely disagree) to 5 (completely agree). The sum of ratings across all 4 items ranges from 4 to 20, where higher scores indicate greater feasibility, and lower scores indicate lower feasibility.
Time Frame: Week 9/Endpoint
Population: Caregivers who completed the FIM. Caregivers responded to the questions for both themselves and their child. Data not collected on staff.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- A+ Treatment Caregiver-Child Dyads: Participants in this arm will be children with ASD and/or ADHD and their caregivers.
  Total participation is expected to require a maximum of 20 weeks (plus optional remote follow-up at 16 week). Diagnostic/screening visits occur between 1 and 6 weeks prior to baseline and start of coaching. Early Start Denver Model (ESDM)-informed parent coaching (~1 hour sessions) is delivered remotely (through telehealth) with a study clinician for 8 weeks and strategies are implemented within the child's typical daily routines by the caregiver. No medication is provided by the study team. Data is collected weekly and final assessment will be obtained at 16 weeks after baseline.
  P-ESDM informed caregiver coaching: Caregiver coaching informed by P-ESDM done remotely (via telehealth)
Arm/Group | A+ Treatment Caregiver-Child Dyads
Number analyzed (Participants) | 19
score on a scale | 18.58 (1.98)

3. Primary Outcome: Acceptability of Intervention (as Measured by the Acceptability of Intervention Measure, AIM)
Description: The AIM is a four-item implementation outcome measure that measures the extent to which a new treatment, or an innovation, can be successfully used or carried out within a given agency or setting. Each item is rated on a 5-point ordinal scale from 1 (completely disagree) to 5 (completely agree). The sum of ratings across all 4 items ranges from 4 to 20, where higher scores indicate greater acceptability, and lower scores indicate lower acceptability.
Time Frame: Week 9/Endpoint
Population: Caregivers who completed the AIM. Caregivers responded to the questions for both themselves and their child. Data not collected on staff.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A+ Treatment Caregiver-Child Dyads
Number analyzed (Participants) | 19
score on a scale | 18.68 (1.73)

4. Primary Outcome: Appropriateness of Intervention (as Measured by the Intervention Appropriateness Measure, IAM)
Description: The IAM is a four-item implementation outcome measure that measures the extent to which a new treatment, or an innovation, can be successfully used or carried out within a given agency or setting. Each item is rated on a 5-point ordinal scale from 1 (completely disagree) to 5 (completely agree). The sum of ratings across all 4 items ranges from 4 to 20, where higher scores indicate greater appropriateness, and lower scores indicate lower appropriateness.
Time Frame: Week 9/Endpoint
Population: Caregivers who completed the IAM. Caregivers responded to the questions for both themselves and their child. Data not collected on staff.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A+ Treatment Caregiver-Child Dyads
Number analyzed (Participants) | 19
score on a scale | 18.21 (2.66)

5. Primary Outcome: Changes From Baseline (Pre-intervention) to Week 9 (Post-intervention) in Fidelity of Intervention Delivery Using an Adapted Version of the Parent Early Start Denver Model (P-ESDM) Caregiver Fidelity Rating System
Description: The caregiver fidelity rating system measure assesses fidelity of the caregiver in using ESDM principles during a joint activity with their child using ratings of performance on 13 items (1-5 scale). The sum of ratings is used for a total score, ranging from 13 to 65, where higher score is greater fidelity and lower scores indicate lower fidelity.
Time Frame: Baseline, Week 9
Population: Caregiver-child dyads who completed the study. Caregivers responded to the questions for both themselves and their child. Data not collected on staff.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | A+ Treatment Caregiver-Child Dyads
Number analyzed (Participants) | 24
score on a scale | 3.75 [1.27 to 6.22]
Statistical Analysis 1: Comparison: A+ Treatment Caregiver-Child Dyads; Within group pre- and post-intervention; Test type: Superiority; p = 0.0047, t-test, 2 sided; Mean Difference (Net) = 3.75, 95% CI 2-sided [1.27 to 6.22], Standard Deviation 5.86

6. Secondary Outcome: Changes From Baseline (Pre-intervention) to 9-weeks (Post-intervention) in Caregiver Sense of Competence Measured by the Parent Sense of Competence Scale.
Description: The parent sense of competence scale is a self-report measure that assesses parenting sense of competence in 3- to 17-year-old children. It is a 16-item 6-point Likert scale questionnaire with ratings ranging from strongly agree (1) to strongly disagree (6). It includes 2 validated factors: satisfaction (9 items) and efficacy (7 items). The scale ranges from 16 to 96, where higher scores indicate greater competence. Change will be measured using the score at each timepoint.
Time Frame: Baseline, Week 9
Population: Caregivers who completed the Parent Sense of Competence Scale. Data not collected on children or staff.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A+ Treatment Caregiver-Child Dyads - Caregivers
Number analyzed (Participants) | 19
score on a scale | 2.21 (7.9)
Statistical Analysis 1: Comparison: A+ Treatment Caregiver-Child Dyads - Caregivers; Within group pre- and post-intervention; Test type: Superiority; p = 0.2383, t-test, 2 sided; Mean Difference (Net) = 2.21, 95% CI 2-sided [-1.6 to 6.02], Standard Deviation 7.90

7. Secondary Outcome: Change From Baseline (Pre-intervention) to 9 Weeks (Post-intervention) in Child Behaviors as Measured by Joint Engagement Rating Inventory (JERI)
Description: Joint Engagement Rating Inventory (JERI) contains eighteen 7-point Likert scale items that characterized various aspects of joint engagement. The items were designed to span the range of possibilities likely to be observed during interactions with 18- to 30-month-old TD children as well as similarly aged and older children with developmental difficulties, including ASD. Reported is the change in the sum of 4 items from the JERI (Joint Engagement, Attention to Caregiver, Responsiveness to Partner's Communication Bids, Fluency and Connectedness) coded by a trained, reliable coder who is naïve with respect to whether the observation is from baseline our outcome using video-recorded caregiver-child interactions. The score range is 4 to 28, where a higher score indicates a greater amount of the aspect of joint engagement.
Time Frame: Baseline, Week 9
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A+ Treatment Caregiver-Child Dyads
Number analyzed (Participants) | 24
score on a scale | -0.71 (3.58)
Statistical Analysis 1: Comparison: A+ Treatment Caregiver-Child Dyads; Within group pre- and post-intervention; Test type: Superiority; p = 0.3426, t-test, 2 sided; Mean Difference (Net) = -0.71, 95% CI 2-sided [-2.22 to 0.80], Standard Deviation 3.58

ADVERSE EVENTS:
Time Frame: Up to 9 weeks
Description: Adverse Event information was not collected on caregivers or staff.
Arm/Group | A+ Treatment Caregiver-Child Dyads - Caregivers | A+ Treatment Caregiver-Child Dyads - Children | A+ Treatment Staff
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/26 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/26 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 14/26 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A+ Treatment Caregiver-Child Dyads - Caregivers (N=0) | A+ Treatment Caregiver-Child Dyads - Children (N=26) | A+ Treatment Staff (N=0)
Abrasions of extremities (Injury, poisoning and procedural complications) | 0 | 1 | 0
Aggression (Psychiatric disorders) | 0 | 2 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Allergic hypersensitivity (Immune system disorders) | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 3 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0
Disturbance in attention (Psychiatric disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Encopresis (Gastrointestinal disorders) | 0 | 1 | 0
Enuresis (Renal and urinary disorders) | 0 | 1 | 0
Frustration (Psychiatric disorders) | 0 | 2 | 0
Gastrointestinal upset (Gastrointestinal disorders) | 0 | 3 | 0
Gastrointestinal virus (Gastrointestinal disorders) | 0 | 1 | 0
Insomnia (Nervous system disorders) | 0 | 4 | 0
Joint sprain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Learning disability (Nervous system disorders) | 0 | 1 | 0
Mood alterations with depression symptoms (Psychiatric disorders) | 0 | 1 | 0
Motor tic (Nervous system disorders) | 0 | 1 | 0
Nasal discharge (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Obsessive rumination (Psychiatric disorders) | 0 | 1 | 0
Pica (Psychiatric disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 2 | 0
Upper respiratory infection (Infections and infestations) | 0 | 3 | 0
Xerosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT05417607/Prot_SAP_001.pdf
  • Informed Consent Form (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT05417607/ICF_000.pdf